CLINICAL TRIAL: NCT02752971
Title: Surgical Wound Infiltration With Sodium Diclofenac Versus Bupivacaine in the Treatment of Acute Postoperative Pain Following Appendectomy
Brief Title: Wound Infiltration With Sodium Diclofenac vs Bupivacaine for Postoperative Pain Following Appendectomy
Acronym: diclofenac
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Central Dr. Luis Ortega (Other)
Responsible Party: Principal Investigator, Beatriz Arismendi Gómez, Medical Doctor, Hospital Central Dr. Luis Ortega
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Sodium Diclofenac in wounds
Record Dates: First submitted 2016-03-20; First posted 2016-04-27 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Diclofenac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- Bupivacaine (Experimental): A dilution of Bupivacaine 0,25% , 15 ml was infiltrated in surgical wound after close the aponeurosis
  Interventions: Drug: Bupivacaine
- Bupivacaine, sodium diclofenac (Experimental): A dilution of Bupivacaine 0,25% and sodium diclofenac 75 mgr, was infiltrated in surgical wound after close the aponeurosis
  Interventions: Drug: Bupivacaine; Drug: Sodium diclofenac
- Sodium diclofenac (Experimental): A dilution of sodium diclofenac 75 mgrs (3ml) and 12 ml of solution 0,9% was infiltrated in surgical wound after close the aponeurosis
  Interventions: Drug: Sodium diclofenac

INTERVENTIONS:
Drug: Bupivacaine
  Arms: Bupivacaine; Bupivacaine, sodium diclofenac
Drug: Sodium diclofenac
  Arms: Bupivacaine, sodium diclofenac; Sodium diclofenac

SUMMARY:
The infiltration of the surgical wound is an effective strategy for postoperative analgesia. Nonsteroidal antiinflammatories are useful in this way.

Objective: To compare the analgesic effectiveness of diclofenac sodium, bupivacaine or bupivacaine plus diclofenac sodium infiltrating wound appendectomies.

Method: Comparative, double blind, American Society Anesthesiologist classification I-II,18-65años. Group 1 (Bupivacaine n = 14), Group 2 (Diclofenac Sodium n = 14), Group 3 (Bupivacaine + Diclofenac Sodium n = 15). Pain at rest and dynamic, rescue analgesic consumption in Post Anesthesia Care Unit (PACU) and 24 hours after surgery were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* American Society Anesthesiologist I- II
* aged 18 and 65
* both sexes
* patients diagnosed with acute appendicitis operated under general anesthesia

Exclusion Criteria:

* Patients known to any allergy of the drugs used in the study
* Different incision approach Mc Burney
* Some intraoperative surgical complications
* Pregnant patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2015-02; Primary Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
rest and dynamic postoperative pain with visual analogue scale | 24 hours of postoperative period
rescue analgesic consumption | 24 hours of postoperative period
appearance of bowel sounds | 24 hours of postoperative period
  auscultation of bowel sounds
changes in rest and dynamic postoperative pain with visual analogue scale | 24 hours of postoperative pain

SECONDARY OUTCOMES:
number of participants with skin suture removal after 10 days | 10 days of postoperative pain